CLINICAL TRIAL: NCT05730309
Title: Point-of-care Ultrasound and Treatment Disparities for Left Ventricular Hypertrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Robert E. Leet and Clara Guthrie Patterson Trust (Unknown)
Responsible Party: Principal Investigator, Cristiana Baloescu, Assistant Professor, Emergency Medicine, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000034381; 000 (Other: YCTG)
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Left Ventricular Hypertrophy
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Intervention Model Description: From the prospective cohort enrolled in Aim 1, after performing the POCUS study, we will offer subjects with LVH on POCUS the three-element intervention (disclosure regarding presence of LVH, pre-specified discharge instruction and referral). Subjects without LVH on POCUS will receive usual ED care and pre-specified discharge instructions about high blood pressure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility: Disclosure, customized discharge and expedited referral instructions (Experimental): Participants enrolled in the Aim 1 cohort with LVH on POCUS will receive the study intervention consisting of disclosure, counseling with set discharge instructions and expedited referral (communication to existing primary care physician OR referral to follow-up clinic if no existing primary care)
  Interventions: Behavioral: Customized discharge and expedited referral instructions

INTERVENTIONS:
Behavioral: Customized discharge and expedited referral instructions — The intervention for subjects with LVH on research POCUS will consist of three elements: 1) disclosure of presence of LVH to subject, ED team and primary care physician (PCP) (if applicable); 2) educational discharge instructions describing high BP, HTN, LVH, implications for development of cardiovascular disease (such as development of heart failure, stroke), options for treatment (lifestyle, medications) and importance of follow-up; A preliminary version will be refined prior to the start of the trial by feedback from ED physicians and patients. Refinement will target content, phrasing, and literacy level. 3) referral to outpatient care, consisting of one of two options, based on whether the subject has an established PCP. For subjects with existing PCP, the study team will call the office, inform about study participation, LVH findings, and secure a follow-up appointment. For those with no PCP, study team will arrange for follow-up to special clinic.

SUMMARY:
The objective of the proposed project is to quantify the prevalence and disparities of undiagnosed left ventricular hypertrophy (LVH) in Emergency Department (ED) patients with persistently elevated asymptomatic BP, and to measure the effect of disclosure, education, and expedited referral on 3-month outpatient follow-up and treatment rates for ED patients with newly diagnosed LVH by POCUS. Additionally, investigators will create a database of annotated clips for future development of a machine learning algorithm for LVH detection on POCUS.

DETAILED DESCRIPTION:
The rationale for the proposed project is that, through bedside LVH detection, ED POCUS can be leveraged to identify those high-risk patients with asymptomatic hypertension (HTN) and improve disease prevention equity, while also ultimately decrease cardiovascular disease burden. The objective of the proposed project is to evaluate the feasibility and impact of LVH determination by POCUS on ED patients with elevated BP, and to quantify disparities in diagnosis and treatment.

This study has 3 Aims:

Aim 1: To quantify the prevalence and disparities of undiagnosed LVH in ED patients with persistently elevated asymptomatic BP. The investigators will enroll a prospective cohort of ED patients with BP > 140/90mmHg on two measurements who will receive POCUS to assess for LVH. The investigators hypothesize an overall LVH prevalence of at least 30%.

Aim 2: To measure the effect of disclosure, education, and expedited referral on 3-month outpatient follow-up and treatment rates for ED patients with newly diagnosed LVH by POCUS. In a single arm feasibility clinical trial, subjects enrolled in the Aim 1 cohort with LVH on POCUS will receive the study intervention consisting of disclosure, counseling with set discharge instructions and expedited referral (communication to existing primary care physician OR referral to a follow-up clinic if no existing primary care). The investigators hypothesize a 50% follow-up rate and a 40% treatment rate.

Aim 3: To create a database of annotated clips for development of an artificial intelligence (AI) algorithm for LVH detection on POCUS. A collection of annotated clips would support subsequent training, validation, and eventual integration into POCUS technology to facilitate larger scale screening and referral efforts.

Aim 1 will have a prospective observational study design. Aim 2 will occur sequentially based on results of POCUS performed as part of Aim 1. Aim 3 will follow a repository creation protocol utilizing the ultrasound clips obtained during Aim 1.

This study will lay the groundwork for future research to evaluate the impact of interventions informed by LVH assessment by POCUS on hypertension control, referral, and cardiovascular outcomes, as well as effectiveness of implementation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Two blood pressure measurements greater than 140 mmHg systolic and greater than 90 mmHg diastolic on two separate vital sign checks obtained as part of routine ED care

Exclusion Criteria:

* Subjects in extremis or lacking capacity to consent
* Active treatment of hypertension within the last year
* History of/known left ventricular hypertrophy
* Active cardiac disease under the care of a cardiologist within last year
* Suspicion for hypertensive emergency by treating ED physician
* Admission to the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of LVH by POCUS | Day 1
  LVH point prevalence will be determined based on ultrasound measurements of left ventricular wall thickness and/or left ventricular mass, expressed as percentage of total population enrolled in the study.

SECONDARY OUTCOMES:
Prevalence of LVH stratified by race, ethnicity and gender | through the end of the study, approximately 6 months
  Prevalence of LVH stratified by race, ethnicity and gender, if sample size allows this. LVH point prevalence by subgroups will be expressed as percentage of patients meeting LVH criteria of total enrolled population in that subgroup (eg men, women, African American, etc).
Rate of successful follow-up in group of subjects with LVH on POCUS | 3 months post-intervention
  Rate of successful follow-up in group of subjects with LVH on POCUS at 3 months post intervention, expressed as percentage of total subjects with successful follow-ups. Successful follow-up is defined as: a clinic appointment was made (either virtual or in-person) and subject presented to this appointment.
Rate of treatment in group of subjects with LVH on POCUS | 3 months post-intervention
  Rate of treatment in group of subjects with LVH on POCUS at 3 months post intervention. Treatment is defined as new medication prescribed for blood pressure management following the ED visit where enrollment occurred.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No